CLINICAL TRIAL: NCT00379886
Title: Comparison of Thiopental and Propofol as Anaesteticum During ECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ECT-Jan2004-Jan2007
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Last update posted 2007-11-14 (Estimated); Status verified 2007-11

CONDITIONS: Depression
Keywords: ECT; Depression; Anesthiticum; Propofol; Thiopental
MeSH Terms: conditions — Depression

INTERVENTIONS:
Drug: Propofol Thiopental

SUMMARY:
Electroconvulsive therapy is the most effective treatment in severe depression and the effect is related to the generalized seizure induced by the treatment. General anesthesia is used during the treatment. Since only a brief period of unconsciousness is required anesthetics with a rapid recovery profile are used.

Methohexital, a barbiturat, is internationally considered "the golden standard", bot other short-acting anesthetics are used. In Denmark the most frequent used anestheticum for ECT is Thiopental, a barbiturat, but also Propofol, a non-barbiturat, is used in many psychiatric departments.

Several studies have shown that Propofol reduce seizure duration in comparison with barbiturates. So far, no studies have demonstrated any clinical implications of the reduced seiziure duration. However, these studies have included rather few patiens, most have been retrospective, and in the only prospective study conducted, uni-lateral ECT was used.

The aim of this study is to compare the clinical effect of ECT in patients anesthesized with either Propofol or Thiopental. The hypothesis is that the shorter duration of seizures found with Propofol as anestheticum will increase the number of treatments needed to clinial respons. Furthermore we want to study differences in EEG-relate parameters previously shown to have prognostic value. Hospitalized patients with major depression, who is to be treated with ECT, are randomized to anesthizia with either Thiopental or Propofol. They are rated with Hamilton depression scale and BDI before treatment, after six treatments and when treatment is concluded. When treatment is ended the patients are furthermore rated with MMSE to evaluate their degree of cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Major depression, hospitalized

Exclusion Criteria:

* age under 18, allergi to anestheticum, out-clinic patients, ECT because of other diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2003-01; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Number of ECT-treatments required to treat depression
Duration of seizures
Amount of energy required to initiate seizure

SECONDARY OUTCOMES:
EEG-related parameters
Changes in seizure-threshold
Haemodynamic parameters
Cognitive impairment

CONTACTS AND LOCATIONS:
Overall Officials: Martin Balslev Jørgensen, M.D, Principal Investigator — Rigshospitalet, Department of Psychiatry, Copenhagen, Denmark
Locations (1):
- Rigshospitalet, Department of Psychiatry, Blegdamsvej 9, Copenhagen, Denmark